CLINICAL TRIAL: NCT04639648
Title: Nutritional Status Evaluation of Hospitalized Patients With Acute Respiratory Failure and COPD
Status: Completed | Type: Observational
Sponsor: Fondazione Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Luca Di Lazzaro, Physician, Clinical Nutrition and Internal Medicine, Fondazione Fatebenefratelli
Other Study IDs: 1465/CE Lazio 1
Record Dates: First submitted 2020-09-26; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Malnutrition; COPD
MeSH Terms: conditions — Malnutrition; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malnutrition is a comorbidity oftenly seen in COPD patients who have progressive chronic inflammation and severity. The investigators aimed to determine the impact of nutritional status and nutrition-related factors on prolonged length of stay in hospitalized patients with acute respiratory failure and COPD. Nutritional status has been defined as an individual's health condition as it is influenced by the intake and utilization of nutrients (Todhunter, 1970). Nutritional status can be defined by energy balance, body composition and body function, moreover the chronic inflammation and the physical activity have an important role. In the study is used some tools (anthropometry, Nutritional Risk Screening [NRS 2002], food intake, body composition, Fat-Free Mass Index [FFMI], diaphragm ultrasound for evaluating diaphragmatic mobility, blood tests, hand) to define nutritional status. The investigatos'll analyze prevalance of malnutrition in the sample and the correlation of malnutrition with prolonged length of stay in hospitalized patients with acute respiratory failure and COPD.

DETAILED DESCRIPTION:
Introduction:

Chronic obstructive pulmonary disease (COPD) is a lung disease characterized by chronic obstruction of lung airflow that interferes with normal breathing and is not fully reversible. In Italy the disease frequency is growing, our last estimate by National Health Service in the year 2014 shows more than 6 cases on 100 people (6% of the population).

Materials and methods:

* Sample selection: 40 partecipants were enrolled in the Internal Medicine Department of S. Giovanni Calibita Fatebenefratelli Hospital in Rome
* Data collection: anamnesis (sex, age, GOLD classification, active pathologies, length of stay in hospital); Nutritional Risk Screening [NRS 2002]; food Intake: as pergentage of ingesta in the last meal; (MMRC) dyspnea scale.
* Anthropometry parameters: height , body weight, arm circumference, triceps skin fold thickness and Body Mass index was calculated [BMI = weight (Kg) / (stature (m))²]
* Body Composition: bioimpedance analysis (fat free mass, fat mass, phase angle, fat free mass index [height-normalized index of FFM, which is calculated by dividing FFM (in kg) by height (in m2) ]).
* Blood tests: albumin (g/dL), transferrin (mg/dL), prealbumin (mg/dL), lymphocytes /mm3, Retinol-binding protein (mg/dL), PCR (mg/L), NLR (neutrophil-lymphocyte ratio)
* Functional examinations: handgrip
* Diaphragm ultrasound performed during quiet respiration. The right diaphragm is analyzed through the liver window. The transducer is placed in the anterior subcostal region between the mid clavicular and anterior axillary lines. The ultrasound beam should reach the posterior part of the diaphragm. In the B mode view, the diaphragm is identified as an echogenic line between the interface of the lung and liver or spleen. Then, M mode is performed to record diaphragmatic excursion during respiration.

Statistics Demographic and clinical features were summarized with the descriptive statistic (mean, standard deviation, median, interquartile range) for continuous variables and with absolute frequencies and percentage for categorical variables. We used Chi-Square Tests or Fisher's Exact Test (if n < 5) for comparison of percentages. We used the Pearson or Sperman correlation to evaluate the relationship between the continuous variables.

Ethical approval and consent to participate All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional and the national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with acute respiratory failure and COPD

Exclusion Criteria:

* chronic renal failure
* cancer
* cirrhosis
* inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 hospitalized patients with acute respiratory failure and COPD.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Correlation between BMI (Kg/m2) and prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD | Baseline
  BMI is a tool to define nutritional status and its correlation with prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD is useful to understand the role of nutritional status in these patients
Correlation between dynapenia using handgrip strength test (Kg) and prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD | Baseline
  The dynapenia is a tool to define nutritional status and its correlation with prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD is useful to understand the role of nutritional status in these patients
Correlation between fat free mass (Kg) and prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD | Baseline
  Body composition (fat free mass) is a tool to define nutritional status and its correlation with prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD is useful to understand the role of nutritional status in these patients
Correlation between food Intake: as pergentage of ingesta in the last meal and prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD | Baseline
  Food intake is a tool to define nutritional status and its correlation with prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD is useful to understand the role of nutritional status in these patients
Correlation between albumin (g/dL) blood serum level on prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD | Baseline
  Albumin is very influenced by nutritional status and low blood level means that nutritional status is not good
Correlation between arm circumference (cm) and prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD | Baseline
  Arm circumference is muscle mass related and is a tool to define nutritional status and its correlation with prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD is useful to understand the role of nutritional status in these patients
Correlation between tricipital skin fold thickness (mm) and prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD | Baseline
  Tricipital skin fold thickness is a tool to define nutritional status and its correlation with prolonged length of stay (days) in hospitalized patients with acute respiratory failure and COPD is useful to understand the role of nutritional status in these patients

SECONDARY OUTCOMES:
Correlation between diaphragm ultrasound performed during quiet respiration (mm) and BMI (Kg/m2) in hospitalized patients with acute respiratory failure and COPD | Baseline
  BMI is a tool that define nutritional status, the aim is to determinate if diaphragm ultrasound is influenced by nutritional status
Correlation between diaphragm ultrasound performed during quiet respiration (mm) and dynapenia using handgrip strength test (Kg) in hospitalized patients with acute respiratory failure and COPD | Baseline
  The dynapenia is a tool to define nutritional status, the aim is to determinate if diaphragm ultrasound is influenced by nutritional status
Correlation between diaphragm ultrasound performed during quiet respiration (mm) and body composition - fat free mass (Kg) in hospitalized patients with acute respiratory failure and COPD | Baseline
  Body composition (fat free mass) is a tool to define nutritional status, the aim is to determinate if diaphragm ultrasound is influenced by nutritional status
Correlation between diaphragm ultrasound performed during quiet respiration (mm) and food Intake: as pergentage of ingesta in the last meal in hospitalized patients with acute respiratory failure and COPD | Baseline
  Food intake is a tool to define nutritional status, the aim is to determinate if diaphragm ultrasound is influenced by nutritional status
Correlation between diaphragm ultrasound performed during quiet respiration (mm) and arm circumference (cm) in hospitalized patients with acute respiratory failure and COPD | Baseline
  Arm circumference is muscle mass related and is a tool to define nutritional status, the aim is to determinate if diaphragm ultrasound is influenced by nutritional status
Correlation between diaphragm ultrasound performed during quiet respiration (mm) and tricipital skin fold thickness (mm) in hospitalized patients with acute respiratory failure and COPD | Baseline
  Tricipital skin fold thickness is a tool to define nutritional status, the aim is to determinate if diaphragm ultrasound is influenced by nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Dario Manfellotto, MD, Study Director — Fatebenefratelli San Giovanni Calibita Hospital
Locations (1):
- Fatebenefratelli San Giovanni Calibita-Isola Tiberina Hospital, Rome, Lazio, Italy